CLINICAL TRIAL: NCT00952627
Title: Mechanism of the Anti-remodeling Activity of the Over-the-counter Dietary Supplement, Pycnogenol, on Age-dependent Process of Cardiac Fibrosis in Aged Hypertensive Subjects With Echocardiographic Evidence of Grade I/II Diastolic Dysfunction
Brief Title: Effects of Pycnogenol on Cardiac Fibrosis and Diastolic Dysfunction in Aged Hypertensive Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not able to recruit qualified patents
Sponsor: University of Arizona (Other)
Collaborators: Horphag Research (Unknown)
Responsible Party: Principal Investigator, Ronald Watson, Prinicpal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UofAFRS 439130
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Cardiac Fibrosis; Diastolic Dysfunction
Keywords: Cardiac fibrosis; Diastolic dysfunction; Hypertension
MeSH Terms: conditions — Hypertension | interventions — pycnogenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pycnogenol (Experimental): 200 mg/day
  Interventions: Dietary Supplement: Pycnogenol
- Control (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pycnogenol — 50 mg tablet, 200 mg/day, 4 tablets/day
  Arms: Pycnogenol
Dietary Supplement: Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether Pycnogenol, a natural pine bark extract, is effective in modifying the age-dependent process of cardiac fibrosis and diastolic function in aged hypertensive subjects.

DETAILED DESCRIPTION:
Diastolic heart failure without left ventricular systolic dysfunction comprises 30% to 50% of heart failure in clinical practice, and hypertensive heart disease is a major cause of this type of heart failure. The complication of myocardial fibrosis should be avoided in hypertensive heart disease, because increasing ventricular stiffness caused by myocardial fibrosis leads to the development of diastolic dysfunction of the heart. Diastolic dysfunction in patients with prolonged hypertension is often associated with myocardial fibrosis in addition to muscular hypertrophy as a final feature of hypertensive heart disease. The high risk of developing maladaptive cardiac remodeling during hypertension, and failure of pharmacological treatments to limit or even reverse this progressive stiffening of the myocardium, has led to the study of effects of Pycnogenol, a bioflavonoid-rich pine bark extract, with pleiotropic actions on cardiovascular system. Pycnogenol prevents adverse hypertension-induced myocardial remodeling in mice, through modulation of gene expression and activity of enzyme matrix metalloproteinases and their tissue inhibitors, affecting myocardial collagen degradation rate. Despite the mounting evidence suggesting the anti-remodeling effect of Pycnogenol in animal models, the clinical efficacy of Pycnogenol in hypertension-induced diastolic dysfunction is unreported. This leads to our central hypothesis that Pycnogenol reverses the hypertension-induced cardiac fibrosis and diastolic dysfunction in hypertensive patients. Therefore in this clinical investigation, we will investigate the effects of Pycnogenol in modifying hypertension-induced cardiac fibrosis (by measuring the serum markers of myocardial fibrosis and collagen turnover) and diastolic dysfunction (by transthoracic echocardiogram). We expect to improve diastolic function and ameliorate myocardial fibrosis with the nutritional supplement Pycnogenol, by modulation of MMPs and TIMPs enzyme activities.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will consist of ambulatory males and females, 50-75 years of age, of any race, diagnosed with hypertension (diagnosis made over 6 months), and echocardiographic evidence of grade I or II diastolic dysfunction.
* There is no need for standardization of hypertension treatment, as we select only patients who have diastolic dysfunction during treatment.

Exclusion Criteria:

* Unstable angina or myocardial infarction in the past 3 months.
* Biochemical evidence of renal or hepatic failure.
* Severe anemia: defined as hemoglobin level less than 7 g/dL.
* Current cancer or other major illness not associated with the heart.
* Bleeding disorders.
* Taking anticoagulants including low dose aspirin.
* Diabetes.
* Known allergy to Pycnogenol.
* Being pregnant or breastfeeding.
* Systolic blood pressure over 180 mmHg or less than 100 mmHg, and Diastolic blood pressure over 110 mmHg or less than 50 mmHg.
* Current smoking.
* Having breast implants.
* Taking any of the following: birth control products, Diethylstilbestrol, Ephedra, ephedrine, or pseudoephedrine (except where used in prescription products), hormone replacement products, Isotretinoin, any product containing mercury, Phentermine in combination with fenfluramine (including but not limited to Pondimin) or dexfenfluramine (Redux).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
cardiac fibrosis (by measuring the serum markers of myocardial fibrosis and collagen turnover) and diastolic dysfunction (by transthoracic echocardiogram) | at baseline and at 4 months

SECONDARY OUTCOMES:
liver and kidney function tests | at baseline and at 4 months
Immunological measurements including the cytokine profile in serum (interleukin (IL)-4, IL-10, interferon-gamma, C-reactive protein). | baseline and at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald R Watson, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Sarver Heart Center, Tucson, Arizona, United States